CLINICAL TRIAL: NCT03560596
Title: Helping Hypertensive Latinos to Improve Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-02974
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Hypertension
Keywords: Latino
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Risk Latino Patients Adherence Intervention (Experimental): 74 high risk Latinos with uncontrolled hypertension
  Interventions: Behavioral: Adherence Intervention
- High Risk Latinos Usual Care (Active Comparator): 74 high risk Latinos with uncontrolled hypertension
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Adherence Intervention — 9 sessions with bilingual health coaches who will utilize a culturally tailored adherence checklist to identify patients specific medication adherence barriers.
  Arms: High Risk Latino Patients Adherence Intervention
Behavioral: Usual Care — standard hypertension treatment recommendations as determined by PCP
  Arms: High Risk Latinos Usual Care

SUMMARY:
Poor medication adherence is a major contributor to inadequate BP control, and is associated with 125,000 deaths annually. Translation of adherence interventions to community-based primary care practices where majority of Latino patients receive care is non-existent. Thus, the development of tailored interventions targeted at improving medication adherence in the Latino population is needed in order to address the racial disparities in BP control between Latinos and whites. This proposal provides a unique opportunity to address this gap in the literature. Using a randomized control design (RCT), the study will evaluate the effect of a culturally tailored, practice-based intervention on medication adherence in 148 high-risk Latino patients with uncontrolled HTN. To facilitate translation into routine practices, the intervention will be integrated into the clinic's electronic medical record (EMR) system, and will be delivered by trained, bilingual Health Coaches.

DETAILED DESCRIPTION:
Latinos are the fastest growing ethnic group of the U.S. with a growth rate of 43% compared to 23% among whites over the past decade. This increase is four times the nation's 9.7% growth rate, and accounts for more than half of the total U.S. population increase of 27.3 million during this period. This growth is accompanied by a significant increase in cardiovascular disease (CVD)-related morbidity and mortality. Despite increasing trends in the awareness and treatment of hypertension (HTN) among all groups, Latinos have the lowest blood pressure (BP) control rates in the U.S. Although barriers to optimal HTN control such as poor access, and low awareness have been used to explain the disparities in BP control between Latinos and whites, BP control rates remain lower among Latinos who receive treatment compared to whites. This enigma may be explained by the disproportionately poorer adherence to prescribed antihypertensive medications among Latinos compared to whites. Poor medication adherence is a major contributor to inadequate BP control, and is associated with 125,000 deaths annually. Despite over 30 years of research dedicated to understanding adherence behaviors in hypertensive patients, data in Latino patients is scant. More importantly, translation of adherence interventions to community-based primary care practices where majority of Latino patients receive care is non-existent.

ELIGIBILITY:
Inclusion Criteria:

* Have uncontrolled hypertension defined as BP>140/90 mmHg on at least two consecutive visits in the past year (or BP>130/80 mmHg for those with diabetes or kidney disease)
* Framingham Risk Scores (FRS) >20% (or at least one CVD risk factor including hyperlipidemia or diabetes)
* Be taking at least one antihypertensive medication;
* Self-identify as Latino

Exclusion Criteria:

* Refuse or are unable to provide informed consent;
* Currently participate in another hypertension study;
* Have significant psychiatric comorbidity

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2016-06-04 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Rate of Medication Adherence assessed with electronic drug monitoring devices (EMD) | 6 Months
  Adherence will be defined as the number of times the EMD records an opening of the pill bottle cap for each day the patient was in the study.

SECONDARY OUTCOMES:
Self-reported medication adherence | 6 Months
  Self-reported adherence will be measured with a validated tool. Adherence will be defined as the percent adherence between baseline and 6 months B. Blood pressure control
Blood pressure reduction | 6 Months
  Difference between the baseline and systolic and diastolic BP readings at 6 months.
Blood pressure control | 6 months
  Rate of blood pressure control at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Schoenthaler, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Schoenthaler A, de la Calle F, Pitaro M, Lum A, Chaplin W, Mogavero J, Rosal MC. A Systems-Level Approach to Improving Medication Adherence in Hypertensive Latinos: a Randomized Control Trial. J Gen Intern Med. 2020 Jan;35(1):182-189. doi: 10.1007/s11606-019-05419-3. Epub 2019 Oct 17. PMID 31625041